CLINICAL TRIAL: NCT00874861
Title: A Pilot Study to Evaluate the Effects of Vaccinations With HLA-A2-Restricted Glioma Antigen-Peptides in Combination With Poly-ICLC for Adults With Recurrent WHO Grade II Gliomas
Brief Title: HLA-A2-Restricted Glioma Antigen-Peptides Vaccinations With Poly-ICLC for Recurrent WHO Grade II Gliomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ian F. Pollack, M.D. (Other)
Collaborators: Musella Foundation (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ian F. Pollack, M.D., Chief, Pediatric Neurosurgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-135; 1R21CA133859 (NIH)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Astrocytoma; Oligoastrocytoma; Oligodendroglioma
Keywords: cancer; brain; tumor; vaccine
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Neoplasms | interventions — Protein Subunit Vaccines; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine + Poly-ICLC (Experimental): Peptide Vaccine + Poly-ICLC
  Interventions: Biological: Peptide vaccine + Poly-ICLC

INTERVENTIONS:
Biological: Peptide vaccine + Poly-ICLC — Subcutaneously in right or left upper arms with intact draining axillary nodes. Each will be injected to the same location in the same arm as the previous vaccine was administered. In case of no intact axillary lymph nodes as draining nodes, vaccines will be administered in the upper thigh on the same side with intact inguinal lymph nodes.
  Vaccine will be administered on weeks 0,3,6,9,12,15,18 and 21. Poly-ICLC First course(20 mg/kg i.m., up to 1640 µg/injection) will be administered on an outpatient basis in the Clinical & Translational Research Center (CTRC)the day of the first GAA/TT-vaccine and on day 4 after the vaccine. For each of the repeated vaccinations (on Weeks 3,6,9,12,15,18 and 21) poly-ICLC will be administered on day of the vaccine and on day 4 after the vaccine.

SUMMARY:
This is a pilot vaccine study in adults with recurrent WHO Grade II gliomas. The purpose of this study is to test the safety and efficacy of an experimental tumor vaccine made from peptides in combination with the study drug Poly-ICLC.

Poly-ICLC, manufactured by Oncovir, Inc., has already been received and is generally well tolerated by subjects in earlier studies and has been shown to decrease the size of brain tumors in some cases.

The immunological and safety data will be used to decide whether a larger study of clinical efficacy is warranted.

DETAILED DESCRIPTION:
This is a pilot study of a vaccination regime that is designed to efficiently induce anti-tumor T-cell responses in patients with recurrent WHO grade II glioma. The proposed regime combines subcutaneous injections of glioma-associated antigen (GAA)-derived cytotoxic T-lymphocyte (CTL) epitope-peptides with simultaneous intramuscular (i.m.) administration of poly-ICLC.

The overall objective of this pilot study is to collect immunological and safety data that will be used to decide whether a larger study of clinical efficacy is warranted in these patients. All patients on the study will be followed for a minimum of 2 years, so that the actual 2-year overall survival (OS), 6-month and 2-year progression-free survival (PFS) rates can be determined in an exploratory manner.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have recurrent supratentorial WHO grade II astrocytoma, oligoastrocytoma or oligodendroglioma that is histologically confirmed either by the previous biopsy or resection, or at the time of re-operation (re-operation before entry to the current study is allowed; however post-surgery Decadron must be off for at least 4 weeks before administration of the first vaccine). Patients may have received prior external beam radiotherapy and/or chemotherapy. With regard to the prior therapy, patients may have had treatment for no more than 2 prior relapses. Relapse is defined as progression following initial therapy (i.e. radiation +/- chemo if that was used as initial therapy). The intent therefore is that patients may have had 3 prior therapies (initial therapy and treatment for 2 relapses). If the patient had a surgical resection for relapsed disease, and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse.
2. HLA-A2 positive based on flow cytometry.
3. Tumor recurrence is defined by the increase of maximum tumor diameter, based on the axial and/or coronal T2 or FLAIR MR images. Increase of tumor size can be based on comparison with previous scans performed up to prior 3 years to allow assessment of slow-growth of the tumor.
4. Patients must have recovered from the toxic effects of prior therapy: 4 weeks from any investigational agent, 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 4 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Principal Investigator. With regard to previous RT, there must be at least 6 months from the completion of RT (or radiosurgery).
5. Participants must be at least 18 years old. For patients under 18 years old, we have a separate, but similar vaccine study through the Children's Hospital in Pittsburgh.
6. All participants must sign an informed consent document.
7. Participants must have a Karnofsky performance status of > 60 (Appendix I).
8. Documented negative serum HCG for female participants of child-bearing age. Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the peptide-based vaccine and poly-ICLC, breastfeeding should be discontinued if the mother is treated in this study.
9. Participants must be free of systemic infection.
10. Participants with adequate organ function as measured by white blood count ≥ 2500/mm3; lymphocytes ≥ 800/mm3; platelets ≥ 100,000/mm3, hemoglobin ≥ 10.0 g/dL, AST, ALT, GGT, LDH, alkaline phosphatase within 2.5 x upper normal limit, and total bilirubin ≤ 2.0 mg/dL, and serum creatinine within 1.5 X upper limit of normal limit. Coagulation tests PT and PTT have to be within normal limits.

Exclusion Criteria:

1. Presence of gliomatosis cerebri, cranial or spinal leptomeningeal metastatic disease.
2. Even if the initial diagnosis was WHO grade II glioma, if the pathological diagnosis for the recurrent disease demonstrate transformation to higher grade (i.e. WHO grade III or IV) gliomas, patients will be excluded from the eligibility.
3. Concurrent treatment or medications including:

   * Radiation therapy
   * Chemotherapy
   * Interferon
   * Allergy desensitization injections
   * Growth factors
   * Interleukins
   * Any investigational therapeutic medication
4. Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded. Mild arthritis requiring NSAID medications will not be exclusionary.
5. Use of immunosuppressives within 4 weeks prior to study entry or anticipated use of immunosuppressive agents. Dexamethasone, or other corticosteroid medications, if used peri-operative period and/or during radiotherapy, must be tapered and discontinued at least 4 weeks before administration of the first vaccine. Topical corticosteroids and Inhaled steroids are acceptable.
6. Participants who have another cancer diagnosis, except that the following diagnoses will be allowed:

   * squamous cell cancer of the skin without known metastasis
   * basal cell cancer of the skin without known metastasis
   * carcinoma in situ of the breast (DCIS or LCIS)
   * carcinoma in situ of the cervix
   * any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 5 years
7. Participants with known addiction to alcohol or illicit drugs.
8. Because patients with immune deficiency are not expected to respond to this therapy, HIV-positive patients are excluded from the study.
9. Patients who previously participated in UPCI 07-057 are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Both immunological and safety data will serve as bases to decide whether a larger follow-up study is warranted. | 4 years

SECONDARY OUTCOMES:
Clinical response: 6 month and 2-year progression-free survival (PFS) will be evaluated based on serial magnetic resonance imaging (MRI) scans. | 4 years
Tumor tissues for biological correlates: for patients who develop progression, biopsy/resection will be encouraged and analyzed for GAA expression status and infiltration of GAA-specific T-cells | 4

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lieberman, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Hillman Cancer Center (University of Pittsburgh Cancer Institute), Pittsburgh, Pennsylvania, United States